CLINICAL TRIAL: NCT00779961
Title: An Investigation for the Optimal Timing of a Cleft Palate Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, David Fisher, Medical Director and Surgeon, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000010915
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Cleft Palate
Keywords: pediatric; cleft palate; plastic surgery; palatoplasty; pharyngoplasty
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Early Cleft Palate Repair (Age group 6-10 months)
  Interventions: Procedure: Palatoplasty
- Group B (Active Comparator): Sick Kids Routine cleft palate repair (age group 10-14 months)
  Interventions: Procedure: Palatoplasty

INTERVENTIONS:
Procedure: Palatoplasty — Routine palatoplasty will be performed under the supervision of one of five surgeons within the Division of Plastic Surgery at Sick Kids
  Arms: Group A
Procedure: Palatoplasty — Palatoplasty will be performed under the supervision of one of five surgeons within the Division of Plastic Surgery at Sick Kids
  Arms: Group B

SUMMARY:
The effect of timing of cleft palate repair on speech development, velopharyngeal functioning, and facial growth remains unknown. The objective of this study is to determine the effectiveness of early palatal repair versus The Hospital for Sick Children (SickKids) routine palatal repair in isolated cleft palate patients by comparing speech development, velopharyngeal functioning and facial growth outcomes. The null hypothesis is no difference in speech development, velopharyngeal functioning and facial growth between early palatal repair and SickKids routine palatal repair in isolated cleft palate patients.

DETAILED DESCRIPTION:
The goals of palatoplasty are to provide an intact palate and to create a normally functioning velopharyngeal mechanism as early as possible without hazard to other aspects of health and development. Two major criteria by which the success of cleft palate surgery is determined are subsequent speech development and facial growth. Therefore, the debate about timing of cleft palate surgery is focused on the need for early palatoplasty for speech purposes versus later palatoplasty to ensure undisturbed facial growth. A compromise solution to this controversy was proposed by Schweckendiek; the soft palate is repaired at an early age leaving the hard palate cleft unrepaired until later in life. The premise is that primary veloplasty will result in a functioning velopharyngeal mechanism for early speech development, while the unrepaired hard palate will allow unrestricted maxillary growth. The speech outcomes of patients who have undergone delayed stage palate repair have been addressed in several studies and case series. However, there is little evidence to support the benefits of delayed stage repair with respect to facial growth and speech development. Results from published studies have shown the speech results to be relatively poor and fistula rates as unacceptably high. These results have lead a vast majority of North American surgeons to favour primary one-stage repair. Yet, the optimum timing of primary palate repair remains unknown. No randomized control trials or prospective cohort studies have been conducted to address this question.

ELIGIBILITY:
Inclusion Criteria:

* Infant diagnosed with non-syndromic isolated unrepaired cleft involving the secondary palate.
* Between newborn and 5 months of age (pre-palate surgical assessment/ consultation.
* Treated at SickKids.

Exclusion Criteria:

* If they are non-Ontario residents;
* If they have clinical features suggestive of an associated syndrome and/or an associated syndrome;
* If they have Pierre Robin sequence;
* If the palate repair cannot be performed before 15 months of age;
* If the extent of clefting is limited to the primary palate or submucous cleft of the soft palate;
* If the child have a combined cleft lip and palate diagnosis

Ages: 1 Day to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2008-04; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be determined by the presence/absence of Velopharyngeal Insufficiency (VPI) at 5 years of age. | 5 years

SECONDARY OUTCOMES:
Surgical Complications: Surgical complications (i.e. fistula and dehiscence) will be evaluated between 6-8 weeks post-operatively and recorded. | 6-8 weeks post-op
Feeding Assessment: A feeding assessment will be conducted pre-surgery (5 months of age) and post surgery (6-8 weeks post-operatively). | 6-8 weeks post-op
Dental and Facial Growth Disturbances measured in patients with isolated secondary plate cleft by analysis of the severity of their malocclusion,and performing a lateral cephalometric analysis | 5 years of age, 11-13 years of age

CONTACTS AND LOCATIONS:
Overall Officials: David M Fisher, MD, FRCSC, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada